CLINICAL TRIAL: NCT03464669
Title: Impacts of Online and Group Perinatal Education: Towards and Optimization of Services
Brief Title: Impacts of Online and Group Perinatal Education
Status: Completed | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHE-148163
Record Dates: First submitted 2018-02-16; First posted 2018-03-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pregnant Women and Partners
MeSH Terms: interventions — Prenatal Education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group prenatal education: Prenatal education delivered in-person by health and social services centers
  Interventions: Other: Prenatal education
- Online prenatal education: Online prenatal education provided or recommended by health and social services centers
  Interventions: Other: Prenatal education
- Control group: Absence of prenatal education

INTERVENTIONS:
Other: Prenatal education — Observational study : natural distribution of participants between groups
  Groups: Group prenatal education; Online prenatal education

SUMMARY:
This project aims to evaluate the impacts of group prenatal education and online prenatal education on health determinants and users' health status.

DETAILED DESCRIPTION:
Prenatal education is a core component of perinatal care and services provided by health institutions. Whereas group prenatal education is the most common educational model, some health institutions have opted to implement online prenatal education to address accessibility issues as well as the evolving needs of future parents. This prospective cohort study aims to evaluate the impacts of group prenatal education and online prenatal education on health determinants and the perinatal health status of parents. It is part of a larger multipronged study using mixed methods.

ELIGIBILITY:
Inclusion Criteria for pregnant women:

* 10-20 weeks of pregnancy
* Living within the targeted geographic territories
* Fluent in French
* Have not given birth previously

Inclusion criteria for partners:

* Partner of pregnant women between 10 and 20 weeks of pregnancy
* Living within the targeted geographic territories
* Fluent in French

Exclusion Criteria:

* Men and women not fulfilling inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women and partners.
  Recruitment methods :
  * By the research team in hospital waiting rooms, before ultrasound appointments
  * By health professionals in community centers during routine appointments
  * Posters with the team's contact information
  * Registration using advertisements on Facebook
Sampling Method: Non-Probability Sample
Enrollment: 1208 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Perinatal Knowledge | 10-20 weeks of pregnancy; 33 weeks of pregnancy
  Measured with an adapted version of the Health Pregnancies Knowledge Survey

SECONDARY OUTCOMES:
Change from Baseline Psychological Distress | 10-20 weeks of pregnancy; 33 weeks of pregnancy; 6 weeks after child birth
  Measured with a validated French version of the 12-item General Health Questionnaire
Change from Baseline Breastfeeding Self-Efficacy | 10-20 weeks of pregnancy; 33 weeks of pregnancy; 6 weeks after child birth
  Assessed with a French version of the Breastfeeding Self-Efficacy Scale Short-Form
Change from Baseline Anxiety | 10-20 weeks of pregnancy; 33 weeks of pregnancy; 6 weeks after child birth
  Assessed with a validated French version of the State-Trait Anxiety Inventory
Change from Baseline Self-Efficacy in the Parenting Role | 10-20 weeks of pregnancy; 33 weeks of pregnancy; 6 weeks after child birth
  Assessed with a French version of the Parent Expectations Survey
Change from Baseline Depression | 10-20 weeks of pregnancy; 33 weeks of pregnancy; 6 weeks after child birth
  Assessed with a French version of the Parent Expectations Survey
Concern about Labour and Birth | 6 weeks after child birth
  Assessed with a French version of the Oxford Worries about Labour Scale
Control during Childbirth | 6 weeks after child birth
  Assessed with a French version of the Labour Agentry Scale
Personal Control in Pain Relief during Childbirth | 6 weeks after child birth
  Assessed with a French version of the Personal Control in Pain Relief Scale
Birth Weight | 6 weeks after child birth
  Self-reported by parents
Personal experience of the COVID-19 crisis and its influence on the use of prenatal education and information services. | 33 weeks of pregnancy; 6 weeks after child birth
  Measured by an in-house questionnaire put together by experts in perinatal care research and in the study of natural disasters and mental health.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No